CLINICAL TRIAL: NCT02605499
Title: Ultra Violet-C Light Evaluation as an Adjunct to Removing Multi-Drug Resistant Organisms (UVCLEAR-MDRO)
Acronym: UVCLEAR-MDRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00063160
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Healthcare Associated Infection; Multidrug Resistant Organisms
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Patient rooms are counted as enrolled since consent was waived and the number of participants is unknown. Total of 83 rooms.
Oversight: Data Monitoring Committee: No

ARMS (2):
- UV-C light disinfection (Experimental): During intervention UV-C light disinfection will be used in hospital patient rooms as an adjunct to routine daily and discharge cleaning.
  Interventions: Other: UV-C light disinfection
- Control (No Intervention): During control period there will be standard discharge and daily room cleaning only, with no UV-C light disinfection.

INTERVENTIONS:
Other: UV-C light disinfection — UV-C light disinfection will be used in hospital patient rooms as an adjunct to routine daily and discharge cleaning.
  Arms: UV-C light disinfection

SUMMARY:
This study examines the impact of UV-C light disinfection as an adjunct to routine daily and discharge patient room cleaning on patient infection and colonization with hospital associated bacteria.

Patient rooms are counted as enrolled since consent was waived and the number of participants is unknown. Total of 83 rooms.

DETAILED DESCRIPTION:
Effective cleaning of the patient environment (the patient room during hospital stay) is subject to human factors and unfortunately is often inconsistent or inadequate. Patient rooms that have residual bacteria after routine environmental cleaning can act as reservoirs for multidrug-resistant organisms (MDROs) and contribute to the spread of MDROs from patient to patient. In the setting of an increased focus on Healthcare-associated Infections such as Clostridium difficile (C. difficile) and multidrug-resistant Gram negative and Gram positive organisms such as carbapenem-resistant Enterobacteriaceae (CRE), vancomycin-resistant Enterococcus (VRE) and methicillin-resistant Staphlococcus aureus (MRSA), Ultra-Violet C (UV-C) light has been shown to be a safe, effective way to decrease the burden of MDROs in patient rooms. However, studies examining the effectiveness of UV-C light when used post daily and discharge patient room cleaning are lacking.

This study is a cluster, randomized, two-period cross over trial to investigate the relationship between environmental decontamination with UV-C light and transmission of VRE and other healthcare-associated bacteria. It investigates the hypothesis that UV-C in addition to daily cleaning leads to decreased patient acquisition of healthcare-associated bacteria.

This study is important to further advance hospital-based infection prevention knowledge of the impact of UV-C light for environmental cleaning.

Patient rooms are counted as enrolled since consent was waived and the number of participants is unknown. Total of 83 rooms.

ELIGIBILITY:
Inclusion Criteria:

* Patient rooms in pre-selected hospital units within Johns Hopkins Hospital

Exclusion Criteria:

* None, intervention is at level of the hospital unit, not the patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Acquisition of Vancomycin Resistant Enterococcus | 2 years
  Rates of Vancomycin Resistant Enterococcus acquisition will be compared between intervention and control periods.
Acquisition of a composite rate of healthcare-associated bacteria: Vancomycin Resistant Enterococcus, Methicillin Resistant Staphylococcus Aureus, hospital-onset bacteremias, Clostridium difficile, and central line associated bloodstream infections. | 2 years
  Rates of Vancomycin Resistant Enterococcus, Methicillin Resistant Staphylococcus Aureus, hospital-onset bacteremias, multidrug resistant gram negative bacteria, Clostridium difficile, and central line associated bloodstream infections will be compared between intervention and control periods.

SECONDARY OUTCOMES:
Acquisition of Vancomycin Resistant Enterococcus (clinical infection) | 2 years
  Rates of Vancomycin Resistant Enterococcus acquisition (clinical infection) will be compared between intervention and control periods.
Acquisition of Vancomycin Resistant Enterococcus (colonization) | 2 years
  Rates of Vancomycin Resistant Enterococcus acquisition (colonization) will be compared between intervention and control periods.
Acquisition of Clostridium difficile (infection) | 2 years
  Rates of Clostridium difficile infection will be compared between intervention and control periods.
Acquisition of Clostridium difficile (colonization or infection) | 2 years
  Rates of Clostridium difficile (colonization or infection) will be compared between the intervention and control arms.
Acquisition of bacteremia | 2 years
  Rates of hospital onset bacteremia will be compared between the intervention and control arms.
Acquisition of Methicillin Resistant Staphylococcus Aureus (clinical) | 2 years
  Rates of Methicillin Resistant Staphylococcus Aureus acquisition (clinical infection) will be compared between intervention and control periods.
Acquisition of Methicillin Resistant Staphylococcus Aureus (colonization) | 2 years
  Rates of Methicillin Resistant Staphylococcus Aureus acquisition (colonization) will be compared between intervention and control periods.
Acquisition of Methicillin Resistant Staphylococcus Aureus (clinical or colonization) | 2 years
  Rates of Methicillin Resistant Staphylococcus Aureus acquisition (clinical or colonization) will be compared between intervention and control periods.
Acquisition of Central line associated bloodstream infections | 2 years
  Rates of Central line associated bloodstream infections in intervention and control arms will be compared.
Acquisition of multidrug resistant gram negative bacteria (colonization) | 2 years
  Rates of multidrug resistant gram negative bacteria acquisition (colonization) will be compared between intervention and control periods.
Acquisition of multidrug resistant gram negative bacteria | 2 years
  Rates of multidrug resistant gram negative bacteria acquisition will be compared between intervention and control periods.
Differences in patient overall satisfaction with hospital stay as assessed by the Hospital Consumer Assessment of Healthcare Providers and Systems Survey. | 2 years
  Patient satisfaction with overall hospital stay will be compared between intervention and control arms.
Differences in patient satisfaction with environmental cleaning as assessed by the Hospital Consumer Assessment of Healthcare Providers and Systems Survey. | 2 years
  Patient satisfaction with environmental cleaning will be compared between intervention and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Maragakis, MD, MPH, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Derived] Rock C, Hsu YJ, Curless MS, Carroll KC, Ross Howard T, Carson KA, Cummings S, Anderson M, Milstone AM, Maragakis LL. Ultraviolet-C Light Evaluation as Adjunct Disinfection to Remove Multidrug-Resistant Organisms. Clin Infect Dis. 2022 Aug 24;75(1):35-40. doi: 10.1093/cid/ciab896. PMID 34636853